CLINICAL TRIAL: NCT05156554
Title: A Multicenter Randomized Controlled Trial of the Efficacy and Safety of PEG-rhG-CSF Compared With rhG-CSF After Autologous Hematopoietic Stem Cell Transplantation for Lymphoma Patients
Brief Title: PEG-rhG-CSF Compared With rhG-CSF in Lymphoma Patients After Autologous Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-ASCT-II-001
Record Dates: First submitted 2021-12-12; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhG-CSF (Experimental): Patients in PEG-rhG-CSF group received PEG-rhG-CSF day+1 after transplantation.
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF (Active Comparator): Patients in rhG-CSF group received rhG-CSF day+1 after transplantation.
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF was given day +1 after autologous stem cell transplantation with a dose of 6mg.
  Arms: PEG-rhG-CSF
Drug: rhG-CSF — rhG-CSF was given day +1 after autologous stem cell transplantation with a dose of 5μg/kg once per day until the count of neutrophil>0.5×10^9 /L.
  Arms: rhG-CSF

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of PEG-rhG-CSF compared with rhG-CSF on the recovery of hematopoietic function after autologous stem cell transplantation in patients with lymphoma.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and safety of PEG-rhG-CSF compared with rhG-CSF in lymphoma patients after autologous hematopoietic stem cell transplantation. Eligible patients were randomly assigned to PEG-rhG-CSF group or rhG-CSF group. Patients in PEG-rhG-CSF group received PEG-rhG-CSF day +1 after transplantation with a dose of 6 mg. Patients in rhG-CSF group received rhG-CSF day +1 after transplantation with a dose of 5μg/kg once per day until the count of neutrophil>0.5×10^9 /L.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 18 and 65 years;
2. hematopoietic stem cell transplantation for the first time;
3. Lymphoma patients with the requirement for autologous;
4. ECOG score ≤2;
5. Estimated survival time > 3 months;
6. All acute toxicity caused by previous chemotherapy or treatment has been restored; 7.1) The absolute value of neutrophils (>1.5×10^9/L); Hemoglobin (> 90 g/L); 2)Upper Limit Normal (ULN) or creatinine clearance rate (>40 mL/min) of serum creatinine (<1.5 times normal value upper limit) (estimated by Cockcroft-Gault formula); Serum total bilirubin < 1.5 times ULN; Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) = 2.5 times ULN; 7) Coagulation function: International Normalized Ratio (INR) = 1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) = 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are using anticoagulant therapy at screening time). Within the expected range; Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (+10%);

8.Not in pregnancy; 9.Written informed consent are acquired.

Exclusion Criteria:

1. Had received autologous hematopoietic stem cell transplantation or allogeneic transplantation;
2. bone marrow involvement;
3. Patients with active autoimmune diseases requiring systematic treatment were excluded according to the clinical judgment of the investigators;
4. Patients with active infections requiring systematic treatment were excluded according to the clinical judgment of the investigators;
5. Serious complications, such as severe infection, heart, lung, liver and kidney dysfunction；
6. patients in fever of unknown origin before medication（>38℃）；
7. central nervous system involvement;
8. Patients that received pelvic radiotherapy;
9. patients will received Chemotherapy or radiotherapy under the diaphragm after transplantation ；
10. Participation or consideration of participation in another biomedical study during the follow-up period of the present trial;
11. Pregnant or lactating women;
12. Serious heart, lung, hemorrhagic disease;
13. Past psychiatric history; incapacitated or restricted;
14. patient's condition increase the risk of receiving the drug treatment or confusion about the toxic reaction；
15. Severe intolerance to the growth factor under study, or hypersensitivity to one of their components;
16. the patients did not comply with the study;
17. Other situation that investigators consider as contra-indication for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Time to neutrophil engraftment | 30 days

SECONDARY OUTCOMES:
The duration of neutrophilic granulocytopenia | 30 days
Incidence of febrile neutrophilic granulocytopenia | 30 days
Time to platelet engraftment and number of platelet transfused to the patient | 30 days
Adverse Event | 30 days
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, professor, Principal Investigator — Sun Yat-sen University